CLINICAL TRIAL: NCT00129467
Title: Methylphenidate for Depressed Cancer Patients in Hospice
Brief Title: Methylphenidate for Depressed Cancer Patients Receiving Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIR 03-194; 01153 (Other: Portland VAMC IRB); 10-0603 (Other: Portland VAMC R&D); CPC-04115-LX (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2013-08

CONDITIONS: Depression; Palliative Care; Cancer; Mental Disorder
Keywords: Depression; Hospice Care; Antidepressive Agents; Methylphenidate; Central Nervous System Stimulant; Pain; Caregiver Burden; Cancer
MeSH Terms: conditions — Depression; Neoplasms; Mental Disorders; Pain; Caregiver Burden | interventions — Methylphenidate; Selective Serotonin Reuptake Inhibitors; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylphenidate + SSRI (Experimental): During the 18-day blind treatment period, subjects will be prescribed methylphenidate 5-10 mg twice per day and selective serotonin reuptake inhibitor (SSRI). Subjects already receiving a SSRI when they begin the study, will continue on the recommended dose of that SSRI; subjects not receiving a SSRI will be prescribed 10-20 mg per day Citalopram. Subjects who respond to methylphenidate treatment will have the option of continuing on methylphenidate, up to 15 mg bid, and an antidepressant in the 6 week open label portion of the study.
  Interventions: Drug: Methylphenidate; Drug: Selective Serotonin Uptake Inhibitor (SSRI)
- Placebo + SSRI (Placebo Comparator): During the 18-day blind treatment period, subjects will be prescribed placebo 1-2 capsules twice per day and selective serotonin reuptake inhibitor (SSRI). Subjects already receiving a SSRI when they begin the study, will continue on the recommended dose of that SSRI; subjects not receiving a SSRI will be prescribed 10-20 mg per day Citalopram.
  Interventions: Drug: Placebo; Drug: Selective Serotonin Uptake Inhibitor (SSRI)

INTERVENTIONS:
Drug: Methylphenidate — Subjects will take methylphenidate 5 mg twice daily (bid) for 3 days, then 10 mg bid for the remainder of the study. Should a subject have a 50% decrease in their depressive symptoms as measured by the Montgomery Asberg Depression Rating Scale (MADRS) at the initial dose of methylphenidate, they will be maintained at that lower dose as long as their MADRS score remains reduced by 50%. During the 18-day blinded treatment period the total daily dose will not exceed 20 mg.
  If subjects have side effects when increasing to 10 mg bid, they will drop back to 5 mg bid. If the participant develops psychosis or cardiac events, they will be discontinued from methylphenidate.
  Subjects who receive methylphenidate and respond with a 50% reduction in MADRS score will have the option to continue in the open label portion of the study for up to 6 weeks. For patients taking methylphenidate 10 mg bid whose MADRS score is > 10 at day 18, the dose may be increased to 15 mg bid.
  Other Names: Ritalin
  Arms: methylphenidate + SSRI
Drug: Placebo — Subjects assigned to placebo will receive 1 capsule of placebo twice per day (bid) for 3 days and then 2 capsules bid for the remainder of the study. Should a subject have a 50% decrease in their depressive symptoms as measured by the Montgomery Asberg Depression Rating Scale (MADRS) at the initial dose of placebo, they will be maintained at that lower dose as long as their MADRS score remains reduced by 50%.
  If subjects have side effects when increasing the dose to 2 capsules bid, they will drop back to 1 capsule bid. If the participant develops psychosis or cardiac events, they will be discontinued from the intervention.
  Arms: Placebo + SSRI
Drug: Selective Serotonin Uptake Inhibitor (SSRI) — Each subject will be treated with a SSRI. Patients who are taking an SSRI at the time of enrollment will continue on the same medication during the 18-day blind treatment period. The prescribed dose will only be adjusted if it is more than the highest dose in the recommended range (fluoxetine to 40 mg, paroxetine to 40 mg, citalopram to 40 mg, sertraline to 150 mg). Patients who are not on a SSRI at the time of enrollment will be prescribed citalopram 10 mg per day for 2 weeks, then 20 mg per day.
  A subject's SSRI may be discontinued if the subject experiences moderate to severe side effects likely attributable to a SSRI. If subjects experience similar symptoms when increasing their citalopram dose to 20 mg per day, they will drop back to 10 mg per day. During the open label extension, the SSRI may be increased, decreased, or changed to a different SSRI or other antidepressant with the exception of venlafaxine and bupropion
  Other Names: Celexa

SUMMARY:
The purpose of this study is to determine whether methylphenidate is an effective treatment for depression and to document the safety and tolerability of methylphenidate in combination with an Selective Serotonin Reuptake Inhibitor (SSRI) in SSRI treated, terminally ill, hospice and palliative care cancer patients. The investigators hypothesize that depressed hospice and palliative care patients will be more likely to have a 50% reduction in scores on a clinical measure of depression after treatment with Methylphenidate plus an SSRI compared to those patients who are taking a placebo plus an SSRI.

DETAILED DESCRIPTION:
Background: Major depressive disorder can be diagnosed in between 5% and 26% of terminally ill patients. This disorder causes suffering, and is associated with suicidality, increased pain, and increased caregiver burden and caregiver depression. Treatment of depression in cancer patients in hospice and palliative care is complicated by shortened life expectancy. Currently-approved antidepressants take several weeks to be effective. Methylphenidate has been reported in case series and very small randomized trials in patients without cancer as a rapidly effective treatment for depression in medically ill patients. There are no randomized controlled trials to test this agent in terminally ill cancer patients.

Objectives: (1) To determine the effectiveness and safety of methylphenidate for depression treatment in cancer patients receiving hospice and palliative care, (2) to explore whether successful treatment of depression is associated with improved quality of life, and (3) to explore whether effective treatment of depression influences caregiver depression and caregiver burden.

Methods: We will conduct an 18-day randomized, double-blind, fixed-dose (10 mg bid), placebo-controlled clinical trial of methylphenidate for depression in eligible veteran and non-veteran cancer patients with advanced cancer in the following settings: inpatient and outpatient hospice, inpatient and outpatient palliative care, and inpatient and outpatient cancer clinics. We will determine whether improvement in depression is mediated by decreased pain and document the safety and tolerability of methylphenidate in these patients. We will explore whether improvement in depression results in improved quality of life for these patients, and decreases caregiver depression and burden.

Eligible patients who answer yes to the question "are you sad or depressed" will be invited to participate. They will complete measures of depression [Structured Clinical Interview for Diagnosis (SCID), Montgomery-Asberg Depression Rating Scale (MADRS) as primary outcome, Hospital Anxiety and Depression Scale (HADS) as secondary outcome], quality of life, pain, and cognition at baseline. MADRS scores must be greater than 19 and SCID positive for depression at study entry. Subjects will be randomized to either methylphenidate plus an SSRI, or placebo plus an SSRI. Subjects may continue any previously prescribed SSRI, or will be prescribed citalopram if untreated. Participants will be evaluated with the same measures as baseline on days 3, 6, 12 and 18 of the study. In an open label portion of the study, methylphenidate-treated patients whose depression has improved will be followed up to 2 months. Cox proportional hazard analysis will be used to analyze the primary outcome. An estimated 104 subjects will be entered over five years. Caregivers will complete measures of depression and caregiver burden at days 0 and 18.

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* Either enrolled in the OHSU radiology/oncology clinic or VA palliative care, and living within 120 miles of the Portland VAMC.
* Life-limiting disease is any type of solid or blood cancer.
* Eighteen years of age or older.
* Life expectancy of 1 year or less as reflected by hospice admission or palliative care status. Although exact life expectancy can not be predicted, actively dying patients with estimated life expectancy of < 10 days are unlikely to be enrolled.
* Diagnosis of major depression disorder as determined by the Structured Clinical Interview for Diagnosis (SCID).
* Significant depressive cognitive symptomatology as determined by a MADRS greater than 19.
* Currently taking an SSRI but still depressed enough to meet eligibility criteria or not taking SSRI but depressed enough to start on SSRI.
* Willing and able to give informed consent to participate in this study as demonstrated by the MacArthur Competence Assessment Tool for clinical research.
* Speaks/understands English.
* For patients at home who cannot self-administer medications, has a caregiver who can assist with administering medication.

Exclusion Criteria:

Exclusion:

* Dementia or Delirium as determined by the Short Portable Mental Status Questionnaire (SPMSQ) score of less than 7.
* Diagnosis of delirium as determined by the Confusional Assessment Method (CAM).
* Any of the following Brief Psychiatric Rating Scale (BPRS) items rated 4 -, elated mood, suspiciousness, hallucinations, excitement, distractibility or motor hyperactivity.
* Severe insomnia.
* Severe anxiety.
* Significant suicidal ideation.
* History of current mental disorder in which depressive symptoms occur, but for which psychostimulants are contraindicated (schizophrenia and bipolar disorder will be based on history; active psychotic symptoms on selected BPRS items).
* History of stimulant abuse or other active, severe substance abuse.
* Contraindications to methylphenidate or an SSRI including significant cardiac arrhythmias; uncontrolled, severe hypertension; moderate-severe angina; seizure disorder; severe COPD; use of medications such as Levodopa, monoamine oxidase inhibitors, and lithium; diagnosis of narrow-angle glaucoma; or history of SSRI-induced hyponatremia,.
* Physical symptoms including increased blood pressure (DBP greater than 115, SBP greater than 180), pulse greater than 120, irregular pulse, or chest pain consistent with angina.
* Treatment for depression with a non-SSRI antidepressant including Bupropion and Venlafaxine during protocol.
* Known serum creatinine > 3.0, or severe liver disease as reflected by jaundice or hepatic encephalopathy.
* Unable to swallow pills, however if patient has gastrostomy tube or feeding tube in place the study medicines may be administered by this route. Pills may be poured into food.
* Receiving hospice care in a skilled nursing facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-02; Primary Completion 2009-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda K. Ganzini, MD MPH, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from February 2005 through August 2009. Potential subjects were recruited from: a VA Nursing Skilled Care Unit, VA outpatient oncology and palliative care clinics, a community hospice and oncology and radiation clinics at a university hospital affiliated with a VA medical center.
Pre-assignment Details: Subjects completed screening scales on depression, cognition, and psychiatric symptoms and their medical records were reviewed to confirm eligibility. 47 subjects were enrolled, 12 did not meet criteria, 1 person declined screening after consenting, 2 subjects were randomized but did not receive the intervention (1 withdrew and 1 became ineligible)
Groups:
- Methylphenidate + SSRI: During the 18-day blind treatment period, subjects will be prescribed Methylphenidate 5-10 mg twice per day and Selective Serotonin Reuptake Inhibitor. Subjects receiving a SSRI when they begin the study, will continue on the recommended dose of that SSRI; subjects not already receiving a SSRI will be prescribed 10-20 mg per day Citalopram. Subjects who respond to methylphenidate treatment will have the option of continuing on methylphenidate, up to 15 mg bid, and an antidepressant in the 6 week open label portion of the study.
- Placebo + SSRI: During the 18-day blind treatment period, subjects will be prescribed placebo 1-2 capsules twice per day and Selective Serotonin Reuptake Inhibitor. Subjects receiving a SSRI when they begin the study, will continue on the recommended dose of that SSRI; subjects not already receiving a SSRI will be prescribed 10-20 mg per day Citalopram.
Period: Received Intervention
Arm/Group | Methylphenidate + SSRI | Placebo + SSRI
Started | 15 | 17
Completed | 9 | 13
Not Completed | 6 | 4
Not completed — Death | 1 | 1
Not completed — Cardiac SAE (hypertension) | 1 | 1
Not completed — Delirium | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Nausea | 1 | 0
Not completed — Intolerance to citalopram | 0 | 1
Not completed — Dizzyness, fatigue | 0 | 1
Period: Open Label for SSRI+Methylphenidate Arm
Arm/Group | Methylphenidate + SSRI | Placebo + SSRI
Started | 4 (Eligible if in methylphenidate arm & had 50% reduction in Montgomery-Asberg Depression Rating score) | 0
Completed | 2 | 0
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Delirium | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of baseline participants is the number of subjects who received the intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate + SSRI | Placebo + SSRI | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15) | 66 (13) | 64 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 8 | 17 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
Marital Status [Number; unit: Participants]
  Married | 4 | 7 | 11
  Single | 2 | 1 | 3
  Divorced | 7 | 5 | 12
  Widowed | 2 | 3 | 5
  Partnership | 0 | 1 | 1
Education [Mean (Standard Deviation); unit: Years] | 13.5 (2) | 11.9 (3.3) | 12.7 (2.8)
Type of Cancer [Number; unit: Participants]
  Gastrointestinal | 5 | 7 | 12
  Pulmonary | 2 | 5 | 7
  Urogenital | 0 | 2 | 2
  Breast | 2 | 0 | 2
  Prostate | 1 | 1 | 2
  Neurological | 0 | 0 | 0
  Dermatological | 2 | 1 | 3
  Head and Neck | 3 | 1 | 4
  Hematological | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Days to Remission of Depression
Description: Days to a 50% or greater reduction in initial Montgomery-Asberg Depression Rating Scale (MADRS) score.
Time Frame: 18 Days
Population: The number of participants analyzed is the number of who received the intervention
Measure: Mean (Standard Error); unit: Days
Arm/Group | Methylphenidate + SSRI | Placebo + SSRI
Number analyzed (Participants) | 15 | 17
Days | 10.3 (1.77) | 8.1 (1.31)

ADVERSE EVENTS:
Time Frame: 30 days after participants' last day in study
Arm/Group | Methylphenidate + SSRI | Placebo + SSRI
Serious Adverse Events (participants affected / at risk) | 7/15 | 4/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate + SSRI (N=15) | Placebo + SSRI (N=17)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
New cardiac symptom (Cardiac disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Frequency threshold for reporting nonserious adverse events was not determined at the start of the study, but a % was required to be entered in order to complete the adverse event module

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes